CLINICAL TRIAL: NCT03817450
Title: Daily Mouth Care to Prevent Pneumonia in Nursing Homes: A Systems-Level Approach
Brief Title: Daily Mouth Care to Prevent Pneumonia in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-2072; 4R01HS022298-03 (AHRQ)
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Aging; Nursing Home; Pneumonia
Keywords: Mouth Care
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daily Mouth Care (Experimental): The intervention consists of training in Mouth Care Without a Battle (MCWB) techniques and support in established quality improvement techniques. MCWB is a system-level, evidence based, tested approach to person-centered daily mouth care, which includes tooth-brushing, flossing, care of the gums, and denture care. MCWB provides training to all certified nursing assistants (CNAs) and nursing supervisors, and also supports the designation and specialized training of a CNA to serve as a dedicated, full-time Oral Care Aide (OCA) to provide mouth care to the residents who are at greatest risk for pneumonia and require specialized support to achieve good oral hygiene.
  Interventions: Behavioral: Daily Mouth Care
- Standard Mouth Care (No Intervention): Nursing homes will continue to provide standard mouth care to all residents. Nursing home staff will not receive training or supplies in the control condition.

INTERVENTIONS:
Behavioral: Daily Mouth Care — Nursing assistants will be trained to provide daily mouth care to all residents in nursing homes. Mouth care supplies will also be provided to intervention nursing homes.
  Arms: Daily Mouth Care

SUMMARY:
This project will determine whether an evidence-based, tested, pragmatic, system-level, comprehensive mouth care program provided to nursing home residents can reduce the incidence of pneumonia. It also will examine matters related to implementation, sustainability, and cost. If effective, the investigators expect this program to be widely adopted and sustained, to result in fewer episodes of pneumonia, and to reduce health-care costs.

DETAILED DESCRIPTION:
Each year, almost two million episodes of pneumonia are suffered by nursing home (NH) residents across the United States, resulting in more deaths than from any other infection. Further, NH residents acquire pneumonia at a rate 6-10 times higher than older adults in the community, indicating that characteristics of these individuals and/or the NH settings put them at increased pneumonia risk.

Pneumonia is an inflammatory condition usually initiated by the introduction of bacteria into the lung, such as through aspiration. In aspiration, contents from the mouth, throat, or stomach that are colonized with pathogenic bacteria are inhaled into the lungs. Poor oral hygiene is therefore a critical risk factor for pneumonia because it increases the volume and infectious nature of secretions from the mouth and throat.

Considering the high rate of pneumonia in NHs and its relationship to oral hygiene, it should come as no surprise that mouth care provided in NHs is poor. Almost 90% of residents require help with tooth brushing, yet only 16% have their teeth brushed regularly. Reasons for insufficient care include time, other priorities, existing procedures, perceptions that oral health is not vital to overall health, and fear of resistant residents.

Evidence is emerging that improved oral care can prevent pneumonia. However, no studies have developed and tested a program designed specifically for widespread adoption and sustainability. Our research team developed the Mouth Care Without a Battle (MCWB) program, and in pilot-testing, MCWB significantly improved tooth brushing and flossing, reduced dental plaque and gingivitis (which harbor the bacteria that can cause pneumonia), and increased staff knowledge and attitudes related to mouth care.

If MCWB is effective in reducing pneumonia and related hospitalizations and mortality, it would constitute a major advance in disease prevention. Therefore, the aims of this evidence-based, tested, matched-pairs cluster randomized trial are:

1a. Compare the incidence of pneumonia in seven mouth care NHs to the incidence of pneumonia in seven control NHs for two years.

Secondarily:

1b. Compare the case-adjusted incidence of pneumonia in mouth care NHs to the case-adjusted incidence in control NHs, and evaluate whether the intervention effects for pneumonia incidence are modified by resident-level risk factors for pneumonia.

1c. Examine the relationship between the overall incidence of pneumonia and change in average oral health status, as measured by the plaque and gingival indices of cross-sectional random samples of 60 residents per NH at baseline and at the end of the study.

2. Examine the implementation and sustainability of the mouth care program, including: (a) staff self-efficacy to provide mouth care; (b) frequency of mouth care and related supervision; (c) use of mouth care products; (d) barriers and facilitators to implementation; and (e) cost of the mouth care program.

3. In regard to secondary outcomes of hospitalization and mortality: 3a. Compare differences in hospitalization and mortality rates (pneumonia and all cause) from baseline through two years for mouth care and control NHs.

3b. Assess the likelihood that the intervention is cost-saving, and estimate the cost per hospitalization avoided attributable to the mouth care program.

These aims will be addressed in a two year matched pairs cluster randomized trial will be conducted in seven pairs of NHs; one half of each pair will be randomly assisted to receive the intervention (MCWB), and the other half will be assigned to the control condition.

ELIGIBILITY:
Inclusion Criteria:

* Residents who are at least 21 years of age and who reside in a participating nursing home
* Residents who have natural teeth and/or dentures and do not require prophylactic antibiotics prior to a dental examination
* Staff members who are at least 21 years of age and who work in a participating nursing home and speak English

Exclusion Criteria:

* Residents with no natural teeth or dentures
* Residents who require prophylactic antibiotics prior to a dental examination
* Non-English speaking staff members
* Staff members who do not provide direct care to residents

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1416 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Incidence of pneumonia over time | Collected every four months during the 2 year study
  The total number of diagnosed cases of pneumonia

SECONDARY OUTCOMES:
Incidence of hospitalizations over time | Collected every four months during the 2 year study
  The total number of hospitalizations
Mortality | Collected every four months during the 2 year study
  The total number of deaths that occur in the nursing home
Staff self-efficacy to provide mouth care | Baseline and 24 months
  The measure will be administered to all CNAs (age 21 and older) in the intervention sites at baseline and 24 months, and to all CNAs (age 21 and older) in the control sites at 24 months (to avoid a possible Hawthorne effect from pre-administration). In the intervention sites, the 24-month measure will include a retrospective pre-test that asks respondents to reflect on their initial self-efficacy after having learned what they might not have known that they did not know previously. The self-efficacy measure has 35 items (Cronbach's alpha α=0.74-0.92), scored 1 (strongly disagree) to 4 (strongly agree). An increase in post-score shows higher self-efficacy to provide mouth care.
Frequency of mouth care | Collected during the entire 2 year study
  Daily mouth care will be documented on a simple log developed for the MCWB pilot study, on which the certified nursing assistant will record daily, for each resident, whether mouth care occurred. If mouth care did not occur, a reason is documented.
Number of times mouth care products were used | Collected during the entire 2 year study
  Use of mouth care products will be will be documented whenever a certified nursing assistant indicates on the mouth care log that mouth care was provided.

OTHER OUTCOMES:
Intervention costs | Collected during the entire 2 year study
  In the intervention NHs, costs measured over the two year study period will include the salary of the certified nursing assistants and nurses; staff time for MCWB training, supervision, and quality improvement meetings; time spent providing mouth care; and product costs. In addition, the investigators will track staff turnover. The costs will be added together to determine the total cost of MCWB implementation.
Staff Turnover | Collected during the entire 2 year study
  The total number of staff resignations and terminations during the two-year study period
Change in Plaque Index Score for Long-Term Care (PI-LTC) over time | Baseline and 24 months
  The Plaque Index for Long-Term Care (PI-LTC) is a modification of the Simplified Oral Hygiene Index. It is derived by separately scoring the buccal and lingual surfaces of six sextants in the mouth (left, front, and right regions of the upper and lower jaw), resulting in 12 separate observations for residents with a full set of teeth; sextants not containing teeth do not receive a score. Within each sextant, the tooth surface with the worst plaque is scratched using an explorer and assigned a score (0=no plaque or stain present; 1=soft plaque covering not more than one third of the tooth surface or presence of extrinsic stains without other plaque regardless of surface area covered; 2=soft plaque covering between one third and two thirds of the tooth surface; or 3=soft plaque covering more than two thirds of the exposed tooth surface). PI-LTC scores range from 0-3 and are the average sextant score. Lower scores are better.
Change in Gingival Index Score for Long-Term Care (GI-LTC) over time | Baseline and 24 months
  The Gingival Index for Long-Term Care (GI-LTC) is a modification of the Gingival Index. Within each sextant, the most inflamed gingival surface is identified, swept using an explorer, and assigned a score (0=no inflammation; 1=mild inflammation, slight change in color, little change in texture; 2=moderate inflammation, glazing, redness, edema, and/or hypertrophy; or 3=severe inflammation, marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration). Overall GI-LTC scores range from 0-3 and are the average sextant score. Buccal and lingual surfaces scores also are calculated. Lower scores are better.
Change in Denture Plaque Index Score (DPI) over time | Baseline and 24 months
  The Denture Plaque Index (DPI) is scored by removing the denture, placing it in a bath of disclosing solution for 30 seconds, rinsing it under lukewarm water for 15 seconds, and assigning a score to each of four quadrants (upper and lower, and lingual and buccal) as follows: 0=no plaque, 1=light plaque (1-25% of area covered), 2=moderate plaque (26-50% of area covered), 3=heavy plaque (51-75% of area covered), or 4=very heavy plaque (76-100% of area covered). Lower scores are better.

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl Zimmerman, PhD, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao Y, Liu C, Lin J, Ng L, Needleman I, Walsh T, Li C. Oral care measures for preventing nursing home-acquired pneumonia. Cochrane Database Syst Rev. 2022 Nov 16;11(11):CD012416. doi: 10.1002/14651858.CD012416.pub3. PMID 36383760
- [Derived] Zimmerman S, Sloane PD, Ward K, Wretman CJ, Stearns SC, Poole P, Preisser JS. Effectiveness of a Mouth Care Program Provided by Nursing Home Staff vs Standard Care on Reducing Pneumonia Incidence: A Cluster Randomized Trial. JAMA Netw Open. 2020 Jun 1;3(6):e204321. doi: 10.1001/jamanetworkopen.2020.4321. PMID 32558913